CLINICAL TRIAL: NCT02136771
Title: Styrian Vitamin D Hypertension Trial: A Randomized, Double-blind, Placebo Controlled Trial to Evaluate the Effects of Vitamin D Supplementation on Systolic Ambulatory Blood Pressure in Vitamin D Deficient Hypertensive Patients
Brief Title: Styrian Vitamin D Hypertension Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT no:2009-018125-70; 2009-018125-70 (EudraCT Number)
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Arterial Hypertension; Vitamin D Deficiency
MeSH Terms: conditions — Hypertension; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Active Comparator): The treatment group receives 2,800 IU vitamin D3 per day as oily drops (Oleovit D3; producer: Fresenius Kabi Austria, A-8055 Graz) for 8 weeks
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Oily drops as placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — The treatment group receives 2,800 IU vitamin D3 per day as oily drops (Oleovit D3, producer: Fresenius Kabi Austria, A-8055 Graz) for 8 weeks
  Arms: Vitamin D3
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
In this randomized, double-blind, placebo-controlled trial we plan to enrol 200 vitamin D deficient hypertensive patients. Our main objective is to evaluate whether vitamin D3 supplementation with 2,800 IU daily for 8 weeks has an effect on 24-hour systolic ambulatory blood pressure (ABP) compared to placebo. In addition, we also aim to evaluate whether vitamin D3 supplementation alters 24-hour diastolic ABP, pulse wave velocity, N-terminal-pro-brain natriuretic peptide (NT-pro-BNP), corrected QT interval (Bazett formula), renin, aldosterone, 24-hour urinary albumin excretion, HOMA-IR (HOmeostatic Model Assessment: Insulin Resistance), triglycerides and HDL-cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* 25-hydroxyvitamin D levels below 30 ng/ml (75 nmol/L)
* Arterial hypertension defined according to recent guidelines as an average office blood pressure on at least two occasions of systolic ≥ 140 and/or diastolic ≥ 90 mmHg or a mean 24-hour ABP of systolic ≥ 125 and/or diastolic ≥ 80, or a home blood pressure of systolic ≥ 130 and/or diastolic ≥ 85 or ongoing antihypertensive treatment which was initiated due to arterial hypertension
* Age of ≥ 18 years
* Written informed consent.

Exclusion Criteria:

* Hypercalcemia defined a serum calcium >2.65 mmol/L
* Pregnancy or lactating women
* Drug intake as part of another clinical study
* Acute coronary syndrome or cerebrovascular events in the previous 2 weeks
* Glomerular filtration rate (GFR) according to the MDRD formula < 15 ml/min/1.73m²
* Systolic 24-hour ABP > 160 mm Hg or < 120 mm Hg
* Diastolic 24-hour ABP > 100 mm Hg
* Change of antihypertensive treatment (drugs and/or lifestyle) in the previous 4 weeks or planned changes of antihypertensive treatment during the study
* Any disease with an estimated life expectancy below 1 year
* Any clinically significant acute disease requiring drug treatment
* Chemotherapy or radiation therapy during the study
* Regular intake of more than 880 International Units (IU) vitamin D per day in the last four weeks before study entry or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
24-hour systolic ambulatory blood pressure | 8 weeks

SECONDARY OUTCOMES:
24-hour diastolic ambulatory blood pressure | 8 weeks
N-terminal-pro-brain natriuretic peptide (NT-pro-BNP) | 8 weeks
corrected QT interval (Bazett formula) | 8 weeks
Renin | 8 weeks
  Plasma renin concentration
Aldosterone | 8 weeks
  Plasma aldosterone concentration
24-hour urinary albumin excretion | 8 weeks
HOMA-IR | 8 weeks
  HOMA-IR (HOmeostatic Model Assessment: Insulin Resistance)
Triglycerides | 8 weeks
HDL-cholesterol | 8 weeks
Pulse wave velocity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Pilz, MD, PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Derived] Grubler MR, Zittermann A, Verheyen ND, Trummer C, Theiler-Schwetz V, Keppel MH, Malle O, Richtig G, Gangler S, Bischoff-Ferrari H, Scharnagl H, Meinitzer A, Marz W, Tomaschitz A, Pilz S. Randomized trial of vitamin D versus placebo supplementation on markers of systemic inflammation in hypertensive patients. Nutr Metab Cardiovasc Dis. 2021 Oct 28;31(11):3202-3209. doi: 10.1016/j.numecd.2021.07.028. Epub 2021 Aug 18. PMID 34629245
- [Derived] Grubler MR, Gaksch M, Kienreich K, Verheyen ND, Schmid J, Mullner C, Richtig G, Scharnagl H, Trummer C, Schwetz V, Meinitzer A, Pieske B, Marz W, Tomaschitz A, Pilz S. Effects of Vitamin D3 on asymmetric- and symmetric dimethylarginine in arterial hypertension. J Steroid Biochem Mol Biol. 2018 Jan;175:157-163. doi: 10.1016/j.jsbmb.2016.12.014. Epub 2016 Dec 24. PMID 28027911
- [Derived] Grubler MR, Gaksch M, Kienreich K, Verheyen N, Schmid J, O Hartaigh BW, Richtig G, Scharnagl H, Meinitzer A, Pieske B, Fahrleitner-Pammer A, Marz W, Tomaschitz A, Pilz S. Effects of Vitamin D Supplementation on Plasma Aldosterone and Renin-A Randomized Placebo-Controlled Trial. J Clin Hypertens (Greenwich). 2016 Jul;18(7):608-13. doi: 10.1111/jch.12825. Epub 2016 Apr 21. PMID 27098193
- [Derived] Ernst JB, Tomaschitz A, Grubler MR, Gaksch M, Kienreich K, Verheyen N, Marz W, Pilz S, Zittermann A. Vitamin D Supplementation and Hemoglobin Levels in Hypertensive Patients: A Randomized Controlled Trial. Int J Endocrinol. 2016;2016:6836402. doi: 10.1155/2016/6836402. Epub 2016 Feb 23. PMID 27006655
- [Derived] Pilz S, Gaksch M, Kienreich K, Grubler M, Verheyen N, Fahrleitner-Pammer A, Treiber G, Drechsler C, O Hartaigh B, Obermayer-Pietsch B, Schwetz V, Aberer F, Mader J, Scharnagl H, Meinitzer A, Lerchbaum E, Dekker JM, Zittermann A, Marz W, Tomaschitz A. Effects of vitamin D on blood pressure and cardiovascular risk factors: a randomized controlled trial. Hypertension. 2015 Jun;65(6):1195-201. doi: 10.1161/HYPERTENSIONAHA.115.05319. Epub 2015 Mar 23. PMID 25801871